CLINICAL TRIAL: NCT07077941
Title: Supporting Mothers With Integrative Care by Midwives for Lifelong Empowerment (SMILE): A Randomized Controlled Trial Comparing Midwife-led Integrative and Fragmented Standard Inpatient Postpartum Care Models on Maternal Satisfaction and Transition to Motherhood
Brief Title: Comparing Integrative Midwife-led vs. Fragmented Inpatient Postpartum Care: Impact on Satisfaction and Transition to Motherhood
Acronym: SMILE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Vera Eschenbach, Patient Flow Managerin, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMC_Model
Record Dates: First submitted 2025-07-02; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Maternal Health Services; Infant, Newborn; Postnatal Care; Breast Feeding; Maternal-Child Relations; Postpartum Depression (PPD); Mental Health; Lactation; Breast Feeding, Exclusive; Patient Satisfaction and Experience With Integrative Therapies; Neonatal Jaundice; Maternal Behavior; Body Weight Decreased; Breast Feeding of Healthy Full Term Infants; Lactation Mastitis; Lactation Disorder - Postpartum Condition or Complication; Lactation Disorder With Baby Delivered; Lactation; Insufficient, Partial
Keywords: Postnatal care; inpatient; maternity competence; satisfaction; integrative care; breastfeeding; maternal behavior
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum; Psychological Well-Being; Patient Satisfaction; Jaundice, Neonatal; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing care model - control group (No Intervention): In a nursing care model, mother and child are cared for separately. The general nurse, who works in the postnatal ward, is responsible for all the mother's personal matters, while the paediatric nurse, who works in the nursery, is responsible for the newborn's affairs. She is the contact person for questions about breastfeeding and helps with newborn care, for example. The daily ward round is routinely carried out by a doctor on the ward. The paediatrician checks the child's state of health in the nursery once or twice during the stay.
- Midwife-led or integrative care model - intervention group (Active Comparator): In a midwife-led or integrative form of care, mother and child are cared for together by a midwife. This midwife is the contact person for all matters concerning the mother or the newborn. She is there for all personal, physical and other concerns and supports and helps with all questions relating to the baby, be it questions about breastfeeding or other topics such as newborn care. She also regularly checks the health of mother and child and consults a doctor if necessary. A paediatrician routinely visits the mother's room once or twice to check the child's state of health.
  Interventions: Other: Integrative care

INTERVENTIONS:
Other: Integrative care — Joint care of mother and child by just one healthcare professional
  Arms: Midwife-led or integrative care model - intervention group

SUMMARY:
The goal of this clinical trial is to compare two different forms of postnatal care to find out which is most beneficial for mothers and their children after birth and with which they are most satisfied. One is a nurse-led, seperate model of care and the other is a midwife-led, integrative model of care. Participants are healthy women between the ages of 18 and 50. They gave birth between 36+0 and 42+0 weeks of pregnancy and had a child. The type of birth is not an inclusion or exclusion criteria. Our hypotheses are: i) that maternal satisfaction with care in a midwife-led, integrative care model is higher than in separate maternal and infant care; ii) that a positive postpartum experience leads to earlier and increased maternity competence; iii) that a higher breastfeeding rate at the time of the survey in the fourth month can be achieved through integrative care. Participants will be randomly assigned, after birth of their child, to either the group cared for by a nurse or the group cared for by a midwife.

DETAILED DESCRIPTION:
A randomised controlled longitudinal study with three data collection points is being conducted on two postnatal wards.

All women who give birth during the study period, meet the inclusion criteria, and provide informed consent are randomised after delivery to one of the two postnatal wards using Randomiser software. Allocation is stratified by parity, induction of labour, and mode of delivery.

In control group, mothers and their newborns receive care separately according to the standard model by registered general nurses (DGKP) and paediatric nurses (DKKP). In intervention group, mothers and their newborns receive care together from midwives and nursing staff within the framework of an integrative care model.

Regardless of the care model, clinical parameters for both mother and child are gathered at discharge according to the medical record. Additionally, demographic data of the mother is recorded. The mothers are also asked to complete the initial part of the WOMBPMSQ, the Barkin Index of Maternal Functioning (BIMF), and the Beginning Breastfeeding Survey-Cumulative (BBS-C) questionnaire.

One month after birth, participants receive a QR code via SMS or email, granting access to the second data collection. At this point, information is collected on current and previous breastfeeding practices, as well as the health status of both mother and child. Additionally, the second part of the WOMBPNSQ and the BIMF are completed once again.

The third and final data collection occurs four months after birth. Participants receive another QR code to access the online survey. Questions focus on past, current, and intended breastfeeding practices, as well as the health status of both mother and child. Furthermore, the BIMF and the Edinburgh Postnatal Depression Scale (EPDS) are completed. The study concludes with an open-ended question.

Following the completion of data collection, the two groups will be compared based on the collected data.

The following validated questionnaires were selected for this project:

* WOMen's views of Birth Postnatal Satisfaction Questionnaire (WOMBPNSQ) (Smith, 2011; Panagopoulou, 2018; Norhayati et al., 2021),
* The Beginning Breastfeeding Survey - Cumulative (BBS-C) (Mulder, 2013),
* Barkin Index of Maternal Functioning (BIMF) (Barkin et al., 2010),
* Edinburgh Postnatal Depression Scale (EPDS) (Bergant et al., 1998). The EPDS and BIMF are already available in validated German translations. The WOMBPNSQ and BBS-C will be translated into German, adapted, and validated as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 50 years at the time of delivery
* Classified as "low-risk" by the obstetric team in the delivery room
* Gestational age at birth between 36+0 and 42+0 weeks
* Singleton birth (only one child born)
* Intent to breastfeed
* Consent to participate in the study

Exclusion Criteria:

* Women younger than 18 or older than 50 at the time of delivery
* Classified as "high-risk" by the obstetric team
* Multiple birth (e.g., twins, triplets)
* No intention or ability to breastfeed the newborn

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 784 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Functioning 1a | within 3 days postpartum
  The Barkin Index of Maternal Functioning is a 20-item self-report measure, that rated on a scale from 0 (Strongly Disagree) to 6 (Strongly Agree). The total score ranges from 0 to 120, with a score of 120 representing perfect functioning
Maternal Functioning 1b | Approximately 28 days postpartum
  The Barkin Index of Maternal Functioning is a 20-item self-report measure, that rated on a scale from 0 (Strongly Disagree) to 6 (Strongly Agree). The total score ranges from 0 to 120, with a score of 120 representing perfect functioning
Maternal Functioning 1c | Approximately 120 days postpartum
  The Barkin Index of Maternal Functioning is a 20-item self-report measure, that rated on a scale from 0 (Strongly Disagree) to 6 (Strongly Agree). The total score ranges from 0 to 120, with a score of 120 representing perfect functioning

SECONDARY OUTCOMES:
Effectiveness of breastfeeding | Within 3 days postpartum
  The Beginning Breastfeeding Survey-Cumulative (BBS-C) has 24 items, that rated on a scale from 1 ( Always) to 5 (Never). A possible total score ranging from 24 to 120. Higher total cumulative scores on the BBS-C indicate greater breastfeeding effectiveness for the mother and the newborn.
Maternal satisfaction with postnatal care | Approximately 28 days postpartum
  The WOMen's views of Birth Postnatal Satisfaction Questionnaires (WOMBPNSQ) has 36 items, that rated from 1 (strongly agree) to 7 (strongly disagree). The total score ranges from 36 to 252.
Detecting symptoms of postnatal depression | Approximately 120 days postpartum
  The Edinburgh Postnatal Depression Scale (EPDS) was developed as 10 items instrument, that rated on a scale from 0 to 3 by order of statements. The total score of the scale could be from 0 to 30, where the higher score indicates a higher intensity of depression symptoms.

OTHER OUTCOMES:
Breastfeeding process and exclusive breastfeeding rate 7a | Approximately 28 days postpartum
  They are asked whether they are still breastfeeding, whether they are exclusive breastfeeding, when and what they are feeding and what plans they have for the future
Breastfeeding process and exclusive breastfeeding rate 7b | Approximately 120 days postpartum
  They are asked whether they are still breastfeeding, whether they are exclusive breastfeeding, when and what they are feeding and what plans they have for the future
Progression of neonatal jaundice | Within 3 days postpartum
  Neonatal jaundice and the question of whether it needs to be treated
Weight progression | Within 3 days postpartum
  Onset postpartum weight loss below/above 10%
Self-assessment of the state of health of mother and child 11a | Within 3 days postpartum
  One question. On a scale from 1 (very bad) to 5 (very good).
Self-assessment of the state of health of mother and child 11b | Approximately 28 days postpartum
  One question. On a scale from 1 (very bad) to 5 (very good).
Self-assessment of the state of health of mother and child 11c | Approximately 120 days postpartum
  One question. On a scale from 1 (very bad) to 5 (very good)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja A. Stamm, PhD, Principal Investigator — Institute for Outcomes Research Center for Medical Data Science Medical University of Vienna; Alex Farr, PhD, Study Director — Medical University of Vienna, Dept. of Obstetrics and Gynecology, Division of Feto-Maternal Medicine
Locations (1):
- General Hospital Vienna; Department of Obstetrics and Feto-Maternal Medicine Head of the Department of Gynaecology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No